CLINICAL TRIAL: NCT07091487
Title: Effectiveness of the Diabetes Homeless Medication Support (D-HOMES) Program on Diabetes Management
Acronym: D-HOMES R01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Katherine Vickery (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Katherine Vickery, Primary Investigator, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY2024-849; R01DK139152 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Homelessness; Behavioral Activation
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care/Education Session (Active Comparator): Brief one-on-one diabetes education session provided by a diabetes wellness coach.
  Interventions: Behavioral: Enhanced Usual Care/ Education
- Diabetes Homeless Medication Support (D-HOMES) (Experimental): 10 one-on-one behavioral treatments by a diabetes wellness coach.
  Interventions: Behavioral: Diabetes Homeless Medication Support

INTERVENTIONS:
Behavioral: Diabetes Homeless Medication Support — There will be 10 one-on-one sessions offered within 12 weeks to participants. Sessions will last approximately 30 minutes. During sessions a diabetes wellness coach will use behavioral activation and motivational interviewing to get to know participants and set goals to improve diabetes care. The coach will encourage a focus on medication adherence behaviors and psychologiccal wellness to the extent that participants are willing. The coach will also help with resource and care coordination. The coach will also provide a tailored tool matched to the patient's needs/goals and tailored diabetes education as needed.
  Arms: Diabetes Homeless Medication Support (D-HOMES)
Behavioral: Enhanced Usual Care/ Education — Trained diabetes wellness coaches will provide approximately 15 minutes of instruction about the basic concepts of diabetes. They will use handouts aligned with American Diabetes Association guidelines. They will use the ask-offer-ask method to review these with participants and answer basic questions. Handouts will cover (1) general diabetes knowledge, (2) healthy eating with diabetes, (3) physical activity with diabetes. The coach will also provide a general tool to support medication adherence (e.g. pillbox).
  Arms: Enhanced Usual Care/Education Session

SUMMARY:
The goal of this clinical trial is to learn if the Diabetes Homelessness Medication Support (D-HOMES) wellness coaching model is effective for adults who speak English or Spanish, have Type 2 diabetes with an HbA1c at or above 7.5, and have recently experienced homelessness. Researchers will compare a one-time education session about diabetes to 10 wellness coaching sessions to see if there are differences between the groups' health outcomes. The main questions it aims to answer are:

* Do D-HOMES participants have greater reductions in HbA1c at 3 months than participants who received education?
* Do D-HOMES participants have greater reductions in HbA1c at 6 and 12 months compared to those who received education?
* Do D-HOMES participants have improvements in blood pressure control, quality of life, self-reported psychological wellness, diabetes distress, and diabetes medication adherence and self-management at 3, 6, and 12 months?
* What factors must be considered to make D-HOMES scalable?

Participants will:

* complete 5 assessments including two baseline assessments and follow-ups at months 3,6, and 12
* participate in a one-time education session or 10 weeks of wellness coaching.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 yrs. or older
2. English or Spanish-speaking
3. Recent homelessness by HUD and HHS definitions

   1. Any housing instability in the last 12 mo. (includes supported housing or worry about paying rent)
   2. Significant housing instability in the last 24 mos. (includes any stay in shelter, outside, or places not meant for human habitation)
4. Self-reported diagnosis of type 2 diabetes with A1c >7.5%, later verified in medical record and study lab. test
5. Plan to stay in local area or be reachable by phone for the next 12 months
6. Willingness to work on medication adherence and diabetes self-care

Exclusion Criteria:

1. Inability to provide informed consent (e.g., presence of a legal guardian, prisoners)
2. Active psychosis or intoxication precluding ability to give informed consent
3. Pregnant or lactating people at initial enrollment, determined by specific screening questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c at 3 months | From Baseline 1 to Month 3 assessment
  Measure effectiveness of D-HOMES (10 BA coach sessions over 3 mos.) vs. enhanced usual care ([EUC], a single brief diabetes educational session and referrals) on glycemic control, measured by HbA1c, among people who have recently experienced homelessness

SECONDARY OUTCOMES:
HbA1c at 6 months | Baseline 1 to 6-month assessment
  Effectiveness of D-HOMES (10 BA coach sessions over 3 mos.) vs. enhanced usual care ([EUC], a single brief diabetes educational session and referrals) on glycemic control, measured by HbA1c, at 6 months
HbA1c at 12 months | Baseline 1 to 12-month assessment
  Effectiveness of D-HOMES (10 BA coach sessions over 3 mos.) vs. enhanced usual care ([EUC], a single brief diabetes educational session and referrals) on glycemic control, measured by HbA1c, at 12 months
Diabetes self-care and medication adherence (DSMQ) - 3 months | Baseline 2 to 3-month assessment
  The Diabetes Self-Management Questionnaire (DSMQ) is a brief, comprehensive 16-item self-report instrument designed to assess four subscales -Glucose Management, Dietary Control, Physical Activity, and Health-Care Use - as well as a global measure called the Sum Scale. This tool uses a likert scale of 0-3.
Diabetes self-care and medication adherence (DSMQ) - 6 months | Baseline 2 to 6-month assessment
  The Diabetes Self-Management Questionnaire (DSMQ) is a brief, comprehensive 16-item self-report instrument designed to assess four subscales -Glucose Management, Dietary Control, Physical Activity, and Health-Care Use - as well as a global measure called the Sum Scale. This tool uses a likert scale of 0-3.
Difficulties with diabetes management (PAID-5) at 3 months | Baseline 2 to 3-month assessment
  The PAID-5 is a short, five-item questionnaire used to assess diabetes-related emotional distress. Each item is scored on a scale of 0 to 4. The total score ranges from 0 to 20, with scores of 8 or above indicating diabetes-related distress.
Difficulties with diabetes management (PAID-5) at 6 months | Baseline 2 to 6-month assessment
  The PAID-5 is a short, five-item questionnaire used to assess diabetes-related emotional distress. Each item is scored on a scale of 0 to 4. The total score ranges from 0 to 20, with scores of 8 or above indicating diabetes-related distress.
MHI-5 at 3 months | Baseline 2 through 3-month assessment
  The Mental Health Inventory - Five Item (MHI-5) includes 5 questions about mental health over the past month. Responses are on a likert scale ranging from 1 = all the time to 6 = none of the time. Raw scores range from a minimum of 5 to a maximum of 30, where higher scores indicate better mental health.
MHI-5 at 6 months | Baseline 2 through 6-month assessment
  The Mental Health Inventory - Five Item (MHI-5) includes 5 questions about mental health over the past month. Responses are on a likert scale ranging from 1 = all the time to 6 = none of the time. Raw scores range from a minimum of 5 to a maximum of 30, where higher scores indicate better mental health.
Euro-QoL-5 at 3 months | Baseline 2 to 3-month assessment
  The EuroQuol-5D-5L has 6 questions. 5 of these questions address mobility, self care, usual activities, pain/discomfort, and anxiety/depression. These 5 questions are answered on a likert scale of 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, 5=unable to/extreme problems. The 6th question is a 0-100 scale of overall health. Data is presented as a health state or a 5-digit code representing the 1-5 responses of the 5 questions.
Euro-QoL-5 at 6 months | Baseline 2 to 6-month assessment
  The EuroQuol-5D-5L has 6 questions. 5 of these questions address mobility, self care, usual activities, pain/discomfort, and anxiety/depression. These 5 questions are answered on a likert scale of 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, 5=unable to/extreme problems. The 6th question is a 0-100 scale of overall health. Data is presented as a health state or a 5-digit code representing the 1-5 responses of the 5 questions.
Blood Pressure at 3 months | Baseline 1 to 3-month assessment
  Recorded in systolic/diastolic mmHg
Blood Pressure at 6 months | Baseline 1 to 6-month assessment
  Recorded in systolic/diastolic mmHg
Body Mass Index (BMI) at 3 months | Baseline 1 to 3-month assessment
  Measured as BMI = weight (kg) / height (m)^2
Body Mass Index (BMI) at 6 months | Baseline 1 to 6-month assessment
  Measured as BMI = weight (kg) / height (m)^2

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Vickery, MD, MSc, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States